CLINICAL TRIAL: NCT06592131
Title: First-in-Human Phase-1, Randomised, Double-Blinded, Placebo Controlled Study to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses, As Well As a Food Effect Study, of BF844 When Administered Orally to Healthy Adult Participants
Brief Title: BF844 Safety and Pharmacokinetic Study in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EyeXCel Pty. Ltd. (Other)
Collaborators: Usher iii Initiative (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BF-844-01
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Usher Syndrome Type 3
Keywords: treatment; intervention; healthy volunteers; Usher syndrome type 3
MeSH Terms: conditions — Usher Syndromes

STUDY DESIGN:
Intervention Model Description: This is a first-in-human, single center, randomized, double-blinded, single and multiple ascending doses (SAD and MAD) and food effect Phase I study in healthy adult volunteers (HV).
  The SAD cohorts will consist of five cohorts of eight participants (6 randomized to treatment + 2 randomized to placebo) in each cohort (Total 40 HV). Additional cohorts may be added.
  The food effect (FE) cohort will consist of 12 participants who receive a single dose of BF844 in a cross-over manner. Each participants will receive the same single dose of BF844 under two separate conditions: one after an overnight fast, and the second following a high-fat breakfast 30 minutes prior to dosing.
  The MAD cohorts will consist of 3 cohorts of eight participants (6 randomized to treatment + 2 randomized to placebo) in each cohort (Total 24 HV). The subjects in MAD cohorts will be dosed once daily for 7 consecutive days. Additional cohorts may be added.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Cohort-1 First dose of SAD cohort (6 treatment + 2 placebo) (Experimental): Drug: BF844
  Interventions: Drug: BF844
- Cohort-2 Second dose of SAD cohort (6 treatment + 2 placebo) (Experimental): Drug: BF844
  Interventions: Drug: BF844
- Cohort-3 Third dose of SAD cohort (6 treatment + 2 placebo) (Experimental): Drug: BF844
  Interventions: Drug: BF844
- Cohort-4 Fourth dose of SAD cohort (6 treatment + 2 placebo) (Experimental): Drug: BF844
  Interventions: Drug: BF844
- Cohort-5 Fifth dose of SAD cohort (6 treatment + 2 placebo) (Experimental): Drug: BF844
  Interventions: Drug: BF844
- Cohort-6 Using one of the BF844 doses(with/without food) that were tested in SAD (Experimental): Drug: BF844
  Interventions: Drug: BF844
- Cohort-7 First dose of MAD cohort (6 treatment + 2 placebo) (Experimental): Drug: BF844
  Interventions: Drug: BF844
- Cohort 8 Second dose of MAD cohort (6 treatment + 2 placebo) (Experimental): Drug: BF844
  Interventions: Drug: BF844
- Cohort 9 Third dose of MAD cohort (6 treatment + 2 placebo) (Experimental): Drug: BF844
  Interventions: Drug: BF844

INTERVENTIONS:
Drug: BF844 — BF844, a small molecule developed by Usheriii Initiative to prevent or delay the progressive hearing and vision loss in patients with Usher syndrome type 3.

SUMMARY:
First-in-Human Phase-1 Clinical Trial to Assess Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of Single and Multiple Ascending Doses of BF844 when Administered Orally to Healthy Adult Participants.

DETAILED DESCRIPTION:
This is a first-in-human, single center, randomized, double-blinded, single and multiple ascending doses (SAD and MAD) and food effect Phase I study in healthy adult volunteers (HV).

The SAD cohorts will consist of five cohorts of eight participants (6 randomized to treatment + 2 randomized to placebo) in each cohort (Total 40 HV). Additional cohorts may be added.

The food effect (FE) cohort will consist of 12 participants who receive a single dose of BF844 in a cross-over manner. Each participants will receive the same single dose of BF844 under two separate conditions: one after an overnight fast, and the second following a high-fat breakfast 30 minutes prior to dosing.

The MAD cohorts will consist of 3 cohorts of eight participants (6 randomized to treatment + 2 randomized to placebo) in each cohort (Total 24 HV). The subjects in MAD cohorts will be dosed once daily for 7 consecutive days. Additional cohorts may be added.

For each cohort, all HV subjects will be enrolled at the same site To optimise participants safety, BF844 will be administered in a staggered manner as per protocol .

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (Participants) will be eligible for enrollment in the study only if they meet ALL the following criteria at time of Screening and pre-dosing:

  1. Healthy male or female between the ages of 18 and 45 years (inclusive) at the time of Screening. Healthy status will be determined by the Investigator based on medical history, clinical laboratory results, vital sign and electrocardiogram measurements, and physical examination at screening.
  2. Willingness and ability to give personal signed informed consent and comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
  3. Weight of at least 45 kg and a body mass index (BMI) ≥ 19.0 and ≤ 32.0 kg/m2 at Screening.
  4. Male participants who are non-sterilized and sexually active with a female partner of childbearing potential must agree to use adequate contraception from the signing of informed consent, throughout the duration of the study, and for 90 days after completion of the study. Male participants must use barrier contraception (e.g., condom). In addition to the male participant using a condom, the female partner of childbearing potential must also be using a highly effective form of contraception (hormonal or non-hormonal). The male participant must be advised and agree not to donate sperm during this period.
  5. Female participants of childbearing potential who are sexually active with a non-sterilized male partner must agree to routinely use highly effective contraception from signing of informed consent, throughout the duration of the study, and for 30 days after completion of the study. A highly effective method of contraception for women of childbearing potential is defined as one that has no higher than a 1% failure rate per year. The acceptable methods of contraception are:

Intrauterine device (IUD), Bilateral tubal occlusion, Vasectomised partner (provided that the partner(s) absence of sperm in the ejaculate has been confirmed and documented), and Sexual abstinence (if it is the preferred and usual lifestyle of the participant).

Exclusion Criteria:

Participants meeting ANY of the following criteria at time of Screening and/or pre-dosing will be excluded from enrollment:

1. Any concomitant disease, condition, or treatment that could interfere with the conduct of the study, or that would, in the opinion of the Investigator or Sponsor, pose an unacceptable risk to the participant in the study or interfere with the interpretation of study data.
2. Has received any investigational compound within 30 days or 5 half-lives, whichever is longer, prior to the first dose of study drug.
3. Participant who is a study site employee or who is an immediate family member of a study site employee, (e.g., spouse, parent, child, sibling). Any participant under duress during the consent process.
4. Participant has any clinically significant illness, such as cardiovascular, neurologic, pulmonary, hepatic, renal (estimated or actual GFR less than 90 mL/minute), metabolic, gastrointestinal, urologic, immunologic, endocrine, or psychiatric disease or disorder, or other abnormality, which may affect safety, or potentially confound the study results. It is the responsibility of the Investigator to assess the clinical significance; however, consultation with the Sponsor and/or CRO MM may be warranted.
5. Participant has a known hypersensitivity to any component of the formulation of BF844.
6. Participant has a positive urine result for drugs of abuse (defined as any illicit drug use) at Screening or Check-in (Day -1).
7. Participant who, in the opinion of the Investigator, has a history of excessive alcohol or drug abuse within one year of Screening.
8. Use of or plans to use medications (e.g., S-warfarin, NSAIDs, phenytoin, omeprazole, and clopidogrel) that are significantly metabolized by CYP2C19/ CYP2C9. Additionally, the use of any medications that could have a significant impact on organ function (e.g., barbiturates, omeprazole, and cimetidine). These drugs are prohibited during the study and within 5 half-lives of the individual agent or within 28 days (whichever is longer) prior to enrollment.
9. Use or intended use of prescription or non-prescription medications (including vitamins or supplements) from 7 days prior to dosing or 5 half-lives (whichever is greater), unless the Investigator or medical delegate considers that such use would not significantly impact participant safety or study data.
10. Participant is pregnant or lactating or intending to become pregnant before, during, or within 30 days since the last dose of the study drug; or intending to donate ova during such time.
11. If male, the participant intends to donate sperm during the course of this study or within 90 days after the last dose of the study drug.
12. Participant has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (i.e., a history of malabsorption, any surgical intervention known to impact absorption [e.g., bariatric surgery or bowel resection], esophageal reflux, peptic ulcer disease, erosive esophagitis, or frequent [more than once per week] occurrence of heartburn).
13. Participant has a positive test result for: (i) hepatitis B surface antigen (HBsAg), (ii) hepatitis C virus (HCV) antibody, or (iii) human immunodeficiency virus (HIV) infection at Screening.
14. Participant has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, or nicotine gum) within 28 days prior to Check-in (Day -1). The cotinine test is positive at Screening or Check-in (Day -1) or if the participant is unwilling to abstain from nicotine-containing products throughout the study.
15. Participant has poor peripheral venous access.
16. Participant has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis) or had a transfusion of any blood product within 90 days prior to the first dose of the study drug.
17. Participant has a clinically significant ECG (QTcF ≥; 450 for males and 470 for females) at Screening or Check-in (Day -1). Entry of any participant with an abnormal, but not clinically significant, ECG must be approved, and documented by signature of the Investigator or medical delegate.
18. Participant has a supine blood pressure outside the ranges of ≥ 90 to ≤ 140 mmHg for systolic and ≥ 40 to ≤ 90 mmHg for diastolic. If out of range, an assessment may be repeated once for eligibility determination at Screening and/or Check-in (Day -1).
19. Participant has a resting heart rate outside the range of 40 to 100 bpm (not on ECGs). If out of range, the assessment may be repeated once for eligibility determination at Screening and/or Check-in (Day -1).
20. Participant has abnormal laboratory values at Screening or Check-in (Day -1) that suggest a clinically significant underlying disease or participant has the following lab abnormalities: ALT and/or AST ≥ 1.5x ULN.
21. Participant is unwilling to avoid strenuous exercise up to 48 hours prior to any safety laboratory blood draws.
22. Participant is unwilling to abstain from consuming caffeine and/or xanthene products (e.g., coffee, tea, chocolate, and caffeine-containing sodas) while confined to the CRU.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2025-03-06 (Estimated); Study Completion 2025-09-06 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and tolerability of BF844 when administered orally at ascending single and multiple doses to healthy adult participants. | Baseline and 14 Days
  Percentage of participants who experience at least 1 treatment-emergent adverse event (TEAE).
To determine the safety and tolerability of BF844 when administered orally at ascending single and multiple doses to healthy adult participants. | Baseline and 14 Days
  Percentage of participants who discontinue due to an adverse event (AE).
To determine the safety and tolerability of BF844 when administered orally at ascending single and multiple doses to healthy adult participants. | Baseline and 14 Days
  Percentage of participants who meet the clinically significant criteria for safety laboratory tests at least once post dose.
To determine the safety and tolerability of BF844 when administered orally at ascending single and multiple doses to healthy adult participants. | Baseline and 14 Days
  Percentage of participants who meet the clinically significant criteria for vital sign measurements at least once post dose.
To determine the safety and tolerability of BF844 when administered orally at ascending single and multiple doses to healthy adult participants. | Baseline and 14 Days
  Percentage of participants who meet the clinically significant criteria for safety electrocardiogram (ECG) parameters at least once post dose.
To determine the safety and tolerability of BF844 when administered orally at ascending single and multiple doses to healthy adult participants. | Baseline and 14 Days
  Treatment-emergent hearing, vision, or balance abnormalities, as measured by audiometry, visual acuity, and clinical examination.

SECONDARY OUTCOMES:
To determine the effect of food on the absorption of BF844 when administered as a single oral dose in healthy participants. | Baseline and 24 hours
  Plasma PK parameters of BF844 at the dose level selected for the food effect study:
  t1/2
To determine the PK of BF844 when administered as multiple oral doses at escalating dose levels in healthy participants. | Baseline and 7 days
  Plasma PK parameters of BF844 at each dose level:
  Cmax
To determine the PK of BF844 when administered as multiple oral doses at escalating dose levels in healthy participants. | Baseline and 7 days
  Plasma PK parameters of BF844 at each dose level:
  AUClast
To determine the PK of BF844 when administered as multiple oral doses at escalating dose levels in healthy participants. | Baseline and 7 days
  Plasma PK parameters of BF844 at each dose level:
  AUC∞
To determine the PK of BF844 when administered as multiple oral doses at escalating dose levels in healthy participants. | Baseline and 7 days
  Plasma PK parameters of BF844 at each dose level:
  t1/2
To determine the PK of BF844 when administered as multiple oral doses at escalating dose levels in healthy participants. | Baseline and 7 days
  Urine PK parameters of BF844 at each dose level:
  AUC0-24hrs
To determine the effect of food on the absorption of BF844 when administered as a single oral dose in healthy participants. | Baseline and 24 hours
  Plasma PK parameters of BF844 at the dose level selected for the food effect study:
  Cmax
To determine the effect of food on the absorption of BF844 when administered as a single oral dose in healthy participants. | Baseline and 24 hours
  Plasma PK parameters of BF844 at the dose level selected for the food effect study:
  tmax
To determine the effect of food on the absorption of BF844 when administered as a single oral dose in healthy participants. | Baseline and 24 hours
  Plasma PK parameters of BF844 at the dose level selected for the food effect study:
  AUClast
To determine the effect of food on the absorption of BF844 when administered as a single oral dose in healthy participants. | Baseline and 24 hours
  Plasma PK parameters of BF844 at the dose level selected for the food effect study:
  AUC∞
To determine the PK of BF844 when administered as multiple oral doses at escalating dose levels in healthy participants. | Baseline and 7 days
  Plasma PK parameters of BF844 at each dose level:
  tmax
To determine the PK of BF844 when administered as multiple oral doses at escalating dose levels in healthy participants. | Baseline and 7 days
  Plasma PK parameters of BF844 at each dose level:
  AUCτ
To determine the PK of BF844 when administered as multiple oral doses at escalating dose levels in healthy participants. | Baseline and 7 days
  Urine PK parameters of BF844 at each dose level:
  Accumulation factor

CONTACTS AND LOCATIONS:
Overall Officials: Benedict Tan, MBBS, FRACP, Principal Investigator — Linear Clinical Research
Locations (1):
- Linear Clinical Research, Perth, Australia, Australia

IPD SHARING:
Plan to Share IPD: No
The results of the study will be published without referring to individual participant data or compromising confidentiality.

REFERENCES:
- [Background] Alagramam KN, Gopal SR, Geng R, Chen DH, Nemet I, Lee R, Tian G, Miyagi M, Malagu KF, Lock CJ, Esmieu WR, Owens AP, Lindsay NA, Ouwehand K, Albertus F, Fischer DF, Burli RW, MacLeod AM, Harte WE, Palczewski K, Imanishi Y. A small molecule mitigates hearing loss in a mouse model of Usher syndrome III. Nat Chem Biol. 2016 Jun;12(6):444-51. doi: 10.1038/nchembio.2069. Epub 2016 Apr 25. PMID 27110679